CLINICAL TRIAL: NCT01927055
Title: A Clinical Study of Patients With Symptomatic Neurogenic Orthostatic Hypotension to Assess Sustained Effects of Droxidopa Therapy
Brief Title: A Clinical Study of Patients With Symptomatic NOH to Assess Sustained Effects of Droxidopa Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to potential competition with a post-marketing study requested by FDA
Sponsor: Chelsea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NOH401
Record Dates: First submitted 2013-08-16; First posted 2013-08-22 (Estimated); Results first posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-12

CONDITIONS: Symptomatic Neurogenic Orthostatic Hypotension; Parkinson's Disease; Multiple Systems Atrophy; Pure Autonomic Failure; Dopamine Beta Hydroxylase Deficiency
Keywords: NOH; OH; PD; MSA; PAF; DBH
MeSH Terms: conditions — Parkinson Disease; Pure Autonomic Failure; dopamine beta hydroxylase deficiency | interventions — Droxidopa; Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Droxidopa (Active Comparator): Droxidopa 100 mg, 200 mg, 300 mg
  Interventions: Drug: Droxidopa
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Droxidopa — Droxidopa at 100 mg, 200 mg, 300 mg
  Other Names: L-threo-3,4-dihydroxyphenylserine, L-threo-DOPS, or L-DOPS
  Arms: Droxidopa
Drug: Placebo — Placebo to match droxidopa capsules and strength designations
  Other Names: Mannitol
  Arms: Placebo

SUMMARY:
Evaluate the clinical efficacy and safety of droxidopa versus placebo over a 17 week (maximum) treatment period in patients with symptomatic NOH.

DETAILED DESCRIPTION:
This is a multi-center, multi-national, randomized, parallel-group, placebo-controlled, double-blind study with a 17 week (maximum) treatment period consisting of an initial, open-label dose titration (up to 2 weeks), followed by a washout period (up to 3 weeks), followed by a 12 week treatment period on a stable dose.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 years and older and ambulatory (defined as able to walk at least 10 meters);

  2. Clinical diagnosis of symptomatic orthostatic hypotension associated with Primary Autonomic Failure (PD, MSA and PAF), Dopamine Beta Hydroxylase Deficiency;

  3. At the Baseline visit (Visit 2), patients must demonstrate:
  1. a score of at least 4 or greater on the Orthostatic Hypotension Symptom Assessment (OHSA) Item #1;
  2. a fall of at least 20 mmHg in their systolic blood pressure, within 3 minutes of standing;

     4. Provide written informed consent to participate in the study and understand that they may withdraw their consent at any time without prejudice to their future medical care;

     Exclusion Criteria:
* 1. Score of 23 or lower on the mini-mental state examination (MMSE);

  2. Concomitant use of vasoconstricting agents for the purpose of increasing blood pressure;
  1. Patients taking vasoconstricting agents such as ephedrine, dihydroergotamine, or midodrine must stop taking these drugs at least 2 days or 5 half-lives (whichever is longer) prior to their baseline visit (Visit 2) and throughout the duration of the study;

     3. Known or suspected alcohol or substance abuse within the past 12 months (DSM-IV definition of alcohol or substance abuse);

     4. Women who are pregnant or breastfeeding;

     5. Women of child bearing potential (WOCP) who are not using at least one method of contraception with their partner;

     6. Male patients who are sexually active with a woman of child bearing potential (WOCP) and not using at least one method of contraception;

     7. Untreated closed angle glaucoma;

     8. Diagnosis of hypertension that requires treatment with antihypertensive medications (short-acting antihypertensives to treat nocturnal supine HTN are allowed in this study) Any significant uncontrolled cardiac arrhythmia;

     9. History of myocardial infarction, within the past 2 years;

     10. Current unstable angina;

     11. Congestive heart failure (NYHA Class 3 or 4);

     12. History of cancer within the past 2 years other than a successfully treated, non-metastatic cutaneous squamous cell or basal cell carcinoma or cervical cancer in situ;

     13. Gastrointestinal condition that may affect the absorption of study drug (e.g. ulcerative colitis, gastric bypass);

     14. Any major surgical procedure within 30 days prior to the Baseline visit (Visit 2);

     15. Previously treated with droxidopa within 30 days prior to the Baseline visit (Visit 2);

     16. Currently receiving any other investigational drug or have received an investigational drug within 30 days prior to the Baseline visit (Visit 2);

     17. Any condition or laboratory test result, which in the Investigator's judgment, might result in an increased risk to the patient, or would affect their participation in the study;

     18. The Investigator has the ability to exclude a patient if for any reason they feel the subject is not a good candidate for the study or will not be able to follow study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horacio Kaufmann, M.D., Principal Investigator — NYU Langone Medical Center
Locations (3):
- United States (3):
  - NYU Langone Medical Center, New York, New York
  - Information on additional locations involved in this clinical trial contact Chelsea Therapeutics, Charlotte, North Carolina
  - Wisconsin Institute for Neurology and Sleep Disorders, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 61 patients enrolled in the open-label dose titration, 16 patients discontinued in the open-label period and 45 patients continued on to the randomized double-blind treatment period.
Groups:
- Open-label Titration: Droxidopa 100 mg, 200 mg
  Droxidopa: 100 mg and 200 mg capsules 100, 200, 300, 400, 500, 600mg TID dosing for up to 2 weeks of treatment
- Droxidopa: Droxidopa 100 mg, 200 mg, 300 mg
  Droxidopa: 100 mg, 200 mg and 300 mg capsules 100, 200, 300, 400, 500, 600mg TID dosing for up to 12 weeks of treatment
Period: Open-label
Arm/Group | Open-label Titration | Droxidopa | Placebo
Started | 61 | 0 | 0
Completed | 45 | 0 | 0
Not Completed | 16 | 0 | 0
Not completed — Adverse Event | 6 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Study Stopped | 4 | 0 | 0
Not completed — Supine Hypertension | 4 | 0 | 0
Not completed — Difficulty attending study visits | 1 | 0 | 0
Period: Double-Blind
Arm/Group | Open-label Titration | Droxidopa | Placebo
Started | 0 | 22 | 23
Completed | 0 | 11 | 10
Not Completed | 0 | 11 | 13
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 3
Not completed — Study Stopped | 0 | 7 | 7
Not completed — Supine Hypertension | 0 | 0 | 1
Not completed — Extended Vacation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Open-Label: Patients entered open label droxidopa dose titration, but did not proceed into the randomization phase.
- Placebo: Placebo
  Placebo: Placebo to match droxidopa capsules and strength designations. 100, 200, 300, 400, 500, 600mg TID dosing for up to 12 weeks of treatment
- Total: Total of all reporting groups
Arm/Group | Open-Label | Droxidopa | Placebo | Total
Number analyzed (Participants) | 16 | 22 | 23 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.3 (6.99) | 70.2 (7.08) | 70.8 (9.00) | 70.5 (8.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 7 | 18
  Male | 14 | 13 | 16 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 16 | 21 | 23 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 2 | 4
  White | 13 | 22 | 21 | 56
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 19 | 22 | 53
  Canada | 4 | 3 | 1 | 8
Primary Diagnosis [Number; unit: participants]
  Parkinson's Disease | 14 | 15 | 18 | 47
  Pure Autonomic Failure | 1 | 3 | 3 | 7
  Multiple System Atrophy | 1 | 4 | 2 | 7
  DBH Deficiency | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Dizziness/ Lightheadedness/ Feeling Faint/ or Feeling Like You Might Blackout (OHSA Item 1)
Description: OHSA item 1 scale range: 0 (none) -10 (worst), likert scale. Change: score at end of study minus score at randomization. A positive score indicates worsening during the double-blind randomized phase relative to value at randomization, while a negative score indicates an improvement in symptom severity.
Time Frame: Change from Randomization to Week 1
Population: Patients entering the double-blind, randomized phase and having a visit at week 1 of the double-blind phase were analyzed.
  Study was stopped when only 5% of planned participants had completed the study to prevent competition with FDA mandated post-marketing requirement study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 22 | 20
units on a scale | -1.1 (3.2) | -0.5 (1.8)

ADVERSE EVENTS:
Time Frame: From end of screening to end of study (up to 17 weeks)
Groups:
- Open-label Titration: All patients treated with study drug during dose titration (1-14 days)
Arm/Group | Open-label Titration | Droxidopa | Placebo
Serious Adverse Events (participants affected / at risk) | 3/61 | 1/22 | 3/23
Other Adverse Events (participants affected / at risk) | 17/61 | 7/22 | 5/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Titration (N=61) | Droxidopa (N=22) | Placebo (N=23)
Mental Impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Parkinson's Disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cyclic vomiting syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis, acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Titration (N=61) | Droxidopa (N=22) | Placebo (N=23)
Headache (Nervous system disorders) | 5 (5) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 2 (6) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (5) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was prematurely terminated; the limited sample size precludes meaningful conclusions on the efficacy or safety of droxidopa in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No